CLINICAL TRIAL: NCT07345923
Title: Predictive Value of a Rectal Swab With Detection of Enterobacteria (ESBL-E), Carbapenemases, and High-level Cephalosporinase (HLC) on the Risk of Infections With C3G-resistant Enterobacteria in Intensive Care
Brief Title: Predictive Value of a Rectal Swab With Detection of Enterobacteria (ESBL-E), Carbapenemases, and High-level Cephalosporinase (HLC) on the Risk of Infections With C3G-resistant Enterobacteria
Acronym: SCREEN ICU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9826
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Infections, Enterobacteriaceae
Keywords: Infections, Enterobacteriaceae; Enterobacterial Infections; High-level cephalosporinase; Carbapenemases; C3G-resistant enterobacteria
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the research is to evaluate the value of testing for ESBL carriage by rectal swab to predict the risk of ESBL-producing Enterobacteriaceae infections in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Who have been in medical or surgical intensive care at Strasbourg University Hospitals (between January 1, 2024, and January 1, 2025)
* Who have undergone rectal screening for carriage of ESBL/HLC/carbapenemase-producing Enterobacteriaceae

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone rectal screening for carriage of ESBL/HLC/carbapenemase-producing Enterobacteriaceae
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of a negative rectal swab for the risk of infection with ESBL-producing Enterobacteriaceae | Up to 12 months
  The negative predictive value (NPV) answers the following question:
  When the test is negative, what is the probability that the person will not develop an infection with these resistant bacteria?
  For example:
  * Out of 100 people with a negative smear test,
  * if 95 never develop an infection, then the negative predictive value is 95%.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France